CLINICAL TRIAL: NCT02310516
Title: Prospective Evaluation of the Impact of Pre-operative Device on the Personal Experience of Brain Awake Surgery: Comparative Study, Randomized
Brief Title: Prospective Evaluation of the Impact of Pre-operative Device on the Personal Experience of Brain Awake Surgery
Acronym: EVECHE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2013-39; RC12_3677 (Registry Identifier: APHM)
Record Dates: First submitted 2014-10-14; First posted 2014-12-08 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-08

CONDITIONS: Brain Awake Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient with preoperative device (Experimental): patients undergoing brain awake surgery with adequate explanations which are provided preoperatively. Preoperative device corresponds to a pre/ perioperative coaching involving the provision of a comprehensive information support on the awake surgery (short video and information brochure) and an interview with an operating room nurse
  Interventions: Device: preoperative adequate explanations about awake surgery
- Patient with standard procedure (Active Comparator): patients undergoing brain awake surgery with standard procedure (without adequate explanations)
  Interventions: Other: no preoperative explanation

INTERVENTIONS:
Device: preoperative adequate explanations about awake surgery
  Arms: Patient with preoperative device
Other: no preoperative explanation
  Arms: Patient with standard procedure

SUMMARY:
The brain awake surgery has recently boomed in neurosurgical oncology but also in epilepsy surgery. The goal of awake surgery is to allow a more precise localization of sensorimotor functions, languages and cognitive to better respect them. Indeed, the interindividual anatomo-functional variations, the lack of specificity of functional explorations radiological magnetic or nuclear, as well as the reorganization of the areas involved in these functions (mechanisms of brain plasticity) in epileptic patients or patients with cerebral tumor do not allow to identify them in preoperatively. Brain awake surgery allows an analysis and a precise real-time identification of areas and networks involved in these functions through a direct electrical stimulation (inhibitory or activatory). Thus, this surgical technique has become a gold standard in surgery of brain lesions located in functional areas.

However, although the brain awake surgery has been practiced since many years, the confidentiality of these informations until recent years explains probably that very little data to be available on the personal experience of this procedure by patients. Studies that have analyzed the perception of the patient or the satisfaction of the patient after surgery in awake conditions were retrospective and included few patients. The investigators experience of lived of this surgery that the investigators have developed in the investigators team since over four years is that on the whole awake surgery is well tolerated if adequate explanations are provided preoperatively and if a minimum of preoperative precautions are observed.

Thus, the investigators have decided to develop a preoperative device that could improve personal experience and well-being of patients undergoing this surgical approach.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a low grade glioma targeted for intervention in the awake brain surgery;
* Subject able to complete a self-administered questionnaire;
* Subjects who have signed a written informed consent and agreeing to abide by the instructions of the protocol

Exclusion Criteria:

* Minor, pregnant or lactating women, not affiliated to the social security system;
* Subject severe respiratory failure;
* Subjects treated with antipsychotic (neuroleptic or lithium);
* Subjects with cognitive impairment degenerative previously documented (Alzheimer, dementia other);
* subject active addict;
* Subject with personal psychiatric history;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Perioperative experience evaluated postoperatively using a self-administered questionnaire (EVAN LR) | 6 days
  perioperative experience evaluated postoperatively using a self-administered questionnaire (EVAN LR)

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France